CLINICAL TRIAL: NCT05546502
Title: A Phase III, Observer-Blind, Randomized, Controlled Study of the Safety and Immunogenicity of SARS-CoV-2 Protein Subunit Recombinant Vaccine in Healthy Children Aged 12-17 Years in Indonesia
Brief Title: Safety and Immunogenicity of SARS-CoV-2 Protein Subunit Recombinant Vaccine in Healthy Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Collaborators: Center for Child Health Universitas Gadjah Mada (CCH-PRO UGM (Unknown); Cipto Mangunkusumo Hospital/Department of Child Health, Faculty of Medicine, University of Indonesia, Jakarta (Unknown); Faculty of Medicine, Andalas University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CoV2-Children-0322
Record Dates: First submitted 2022-09-04; First posted 2022-09-19 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Vaccine Reaction; Vaccine Adverse Reaction

STUDY DESIGN:
Intervention Model Description: Vaccine candidate and active comparator are masking
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Vaccine candidate and active comparator are masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 Protein Subunit Recombinant Vaccine (Experimental): 2 doses of COVID-19 Protein Subunit Recombinant Vaccine administered with 28 days interval (0.5 mL per dose)
  Interventions: Biological: SARS-CoV-2 Protein Subunit Recombinant Vaccine
- Active Comparator (Active Comparator): 2 doses of Covovax® - administered with 28 days interval (0.5 mL per dose)
  Interventions: Biological: Active Comparator

INTERVENTIONS:
Biological: SARS-CoV-2 Protein Subunit Recombinant Vaccine — SARS-CoV-2 RBD subunit recombinant protein, manufactured by PT. Bio Farma
  Arms: COVID-19 Protein Subunit Recombinant Vaccine
Biological: Active Comparator — Covovax
  Arms: Active Comparator

SUMMARY:
A Phase III, Observer-blind, randomized, active-controlled prospective intervention study

DETAILED DESCRIPTION:
This trial is randomized, prospective intervention study. A total of 1,050 subjects aged 12-17 years (COVID-19 vaccine naive) who are willing to participate in the study by signing the consent form, will be involved in this trial.

The subjects will be divided into twostudy subsets, namely Main Study and Exploratory Study.

Main Study for immunogenicity and safety evaluation.

Exploratory Study for cellular immunity evaluation,

ELIGIBILITY:
Inclusion Criteria:

1. Clinically healthy children aged 12-17 years.
2. Parent and/or legal guardian has been informed properly regarding the study and signed the informed consent form (and assent for subjects aged 12-17 years).
3. Parent and/or legal guardian will commit to comply with the instructions of the investigator and the schedule of the trial.

Exclusion Criteria:

1. Subjects concomitantly enrolled or scheduled to be enrolled in another trial.
2. History of vaccination with any COVID-19 vaccine (based on anamnesis).
3. Subjects who have history of COVID-19 in the last 3 months (based on anamnesis).
4. Evolving mild, moderate or severe illness, especially infectious disease or fever (body temperature ≥37.5℃, measured with infrared thermometer/thermal gun).
5. History of asthma, history of allergy to vaccines or vaccine ingredients, and severe adverse reactions to vaccines, such as urticaria, dyspnea, and angioneurotic edema.
6. History of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection.
7. Patients with serious chronic diseases (serious cardiovascular diseases, uncontrolled hypertension and diabetes, liver and kidney diseases, malignant tumors, etc) which according to the investigator might interfere with the assessment of the trial objectives.
8. Subjects who have any history of confirmed or suspected immunosuppressive or immunodeficient state, or received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulins, blood-derived products or long-term corticosteroid therapy (> 2 weeks)).
9. Subjects who have history of uncontrolled epilepsy or other progressive neurological disorders, such as Guillain-Barre Syndrome.
10. Subjects receive any vaccination (other than COVID-19 vaccine) within 1 month before and after IP immunization.
11. Female who are pregnant or planning to become pregnant during the study period (judged by self-report of subjects and urine pregnancy test results).

11. Subjects plan to move from the study area before the end of study period.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1050 (Actual)
Dates: Start 2022-10-09 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
To evaluate immunogenic non-inferiority immune response of SARS-CoV-2 neutralizing antibody of Bio Farma vaccine compared to vaccine control at 14 days after primary series | 14 days after primary series
  Geometric Mean Titer (GMT) and GMT ratio of neutralizing antibody to the SARS-CoV-2, measured by neutralization assay (against omicron variant) at 14 days after primary series

SECONDARY OUTCOMES:
To evaluate SARS-CoV-2 (RBD)-binding IgG antibody titer before and 14 days after primary series of Bio Farma vaccine. | 14 days after primary series
  Seroconversion rate and Seropositive rate of neutralizing antibody at baseline and 14 days after primary series vaccination.
To evaluate safety of SARS-CoV-2 Protein Subunit Recombinant Vaccine (Bio Farma). | 28 days after each dose
  Local reactions and systemic events
To evaluate safety of SARS-CoV-2 Protein Subunit Recombinant Vaccine (Bio Farma). | 12 months after primary series
  Serious Adverse Event
To compare safety between SARS-CoV-2 protein subunit recombinant vaccine (Bio Farma) and control group. | 28 days after each dose
  local reactions, systemic events
To compare immunogenicity between SARS-CoV-2 protein subunit recombinant vaccine (Bio Farma) and control group. | 28 days after each dose
  SARS-CoV-2 (RBD)-binding IgG antibody titer, neutralizing antibody
To evaluate antibody persistence 3, 6 and 12 months after primary series | 3, 6 and 12 months after primary series
  SARS-CoV-2 (RBD)-binding IgG antibody titer, neutralizing antibody

CONTACTS AND LOCATIONS:
Overall Officials: Cahya Satria, MD, Principal Investigator — CC PRO UGM; Bernie Medise, MD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia; Asrawati Asrawati, MD, Principal Investigator — Faculty of Medicine Universitas Andalas
Locations (10):
- Indonesia (10):
  - Bali Mandara Hospital, Denpasar, Bali
  - Universitas Udayana Hospital, Denpasar, Bali
  - RSUD Hj. Anna Lasmanah, Banjarnegara, Central Java
  - Abdoel Moeloek Hospital, Bandar Lampung, Lampung
  - Rumpin Primary Health Care, Bogor, West Java
  - Duren Seribu Primary Health Care, Depok, West Java
  - Pasir Putih Primary Health Care, Depok, West Java
  - Universitas Mataram Hospital, Mataram, West Nusa Tenggara
  - M Djamil Hospital, Padang, West Sumatra
  - RS Universitas Andalas, Padang, West Sumatra